CLINICAL TRIAL: NCT02697513
Title: The 'Bekele Afessa Scan-Teach-Treat Approach' to Improve Care of Patients With Acute Infection at the Gitwe Hospital in Gitwe/Rwanda
Brief Title: The 'Bekele Afessa Scan-Teach-Treat Approach'
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Salzburg (Other)
Collaborators: Gitwe Hospital and Gitwe School of Medicine (Unknown); Mayo Clinic (Other); Surviving Sepsis Campaign (Unknown); University of Nebraska Medical (Unknown)
Responsible Party: Principal Investigator, Martin W Duenser, MD, DESA, EDIC, Lt. OA Dr., University of Salzburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01
Record Dates: First submitted 2016-02-14; First posted 2016-03-03 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Infection; Sepsis
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Before Period (No Intervention): Collection of patient-related data without interventions being made
- After Period (Active Comparator): Implementation of a simple infection management protocol as well as a 'Sepsis First Aid' kit to assist in the management of patients with acute infection
  Interventions: Behavioral: simple infection management protocol

INTERVENTIONS:
Behavioral: simple infection management protocol — Implementation of a simple management protocol to improve care of patients with acute infection. Implementation will be assisted by a 1.5-day focused training program.
  Arms: After Period

SUMMARY:
Infection and sepsis are among the leading causes of death worldwide, particularly in middle- and low-income countries.The Surviving Sepsis Campaign has launched an initiative to improve sepsis care in resource-limited settings by employing the 'Scan-Teach-Treat' Approach. In this prospective before-after study, three interventions will be performed: First four months period: collection of baseline data on the clinical management of patients with acute infection. Second four months period: During the first days, a 1.5-day focused training program will be performed (participants: health care workers of primary care facilities within the catchment area of the Gitwe hospital and health care workers of the Gitwe hospital). Then, a simple management protocol to care for patients with an acute infection will be implemented into clinical practice. During the third four months period, a 'Sepsis First Aid' kit containing essential resources to treat patients with an acute infection (antimicrobials, fluids, data documentation sheet) will be distributed to primary care facilities and the emergency department of the Gitwe hospital. During the 8 months following the focused training program (periods 2 and 3), data collection will continue. It is hypothesized that implementation of a simple clinical management protocol and exposure of health care workers in the Gitwe Hospital area to a focused training program on the management of acute infections will increase the rate of evidence-based interventions performed in patients with an acute infection during the first six hours after hospital admission (administration of oxygen and fluids whenever indicated, timely administration of antimicrobial drugs, source control measures).

DETAILED DESCRIPTION:
Infection and sepsis are among the leading causes of death worldwide. The annual burden of infectious diseases is particularly high in middle- and low-income countries. The Surviving Sepsis Campaign released guidelines for severe sepsis and septic shock management, whose implementation improved sepsis outcomes. Despite these benefits, the Surviving Sepsis Campaign cannot be implemented in middle- or low-income countries due to lack of training and resources. This leaves those clinicians caring for the worldwide majority of patients suffering from acute infection without standardized and adoptable guidance for sepsis. The Surviving Sepsis Campaign has launched an initiative to improve sepsis care in resource-limited settings by employing the 'Scan-Teach-Treat' Approach. This approach consists of the following three steps: Step 1 - scanning the region of interest for key elements of regional epidemiology of acute infectious diseases as well as elements of the teach and treat module; Step 2 - implementing a focused training program on the management of acute infectious diseases; Step 3 - implementing a 'Sepsis First Aid kit' into clinical practice.

In this prospective before-after study, this approach will be piloted at the Gitwe Distict Hospital in Gitwe, rural Rwanda. During three four month periods, three interventions are planned: First four months period: collection of baseline data on the clinical management of patients with acute infection. Second four months period: During the first days, a 1.5-day focused training program will be performed (participants: health care workers of primary care facilities within the catchment area of the Gitwe hospital and health care workers of the Gitwe hospital). Then, a simple management protocol to care for patients with an acute infection will be implemented into clinical practice. During the third four months period, a 'Sepsis First Aid' kit containing essential resources to treat patients with an acute infection (antimicrobials, fluids, data documentation sheet) will be distributed to primary care facilities and the emergency department of the Gitwe hospital. During the 8 months following the focused training program (periods 2 and 3), data collection will continue. It is hypothesized that implementation of a simple clinical management protocol and exposure of health care workers in the Gitwe Hospital area to a focused training program on the management of acute infections will increase the rate of evidence-based interventions performed in patients with an acute infection during the first six hours after hospital admission (administration of oxygen and fluids whenever indicated, timely administration of antimicrobial drugs, source control measures). In addition to the main analysis, study endpoints will be analyzed separately for the following á priori defined sub-groups: children (<15 years); patients with malaria; patients positive for HIV; patients referred to from primary health care centers.

ELIGIBILITY:
Inclusion Criteria:

all patients admitted to Gitwe Hospital because of a suspected or confirmed acute infectious disease

Exclusion Criteria:

* age <28 days of life
* known allergy to any study-related drug
* limited therapy due to terminal disease
* refusal of written informed consent

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1594 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of evidence-based interventions performed in study patients during six hours after hospital admission before and after the focused training program and implementation of the clinical management protocol. | Six hours after hospital admission
  Evidenced based interventions are defined as initiation of antimicrobials, surgical source control (if applicable), oxygen administration (in case of respiratory distress) and fluid resuscitation (in case of tissue hypoperfusion)

SECONDARY OUTCOMES:
Prevalence of sepsis | 72 hours after hospital admission
Hospital mortality | 28 days after hospital admission or at hospital discharge
Time to initiation of evidence-based interventions after Hospital admission | Six hours after hospital admission
  Evidenced based interventions are defined as initiation of antimicrobials, surgical source control (if applicable), oxygen administration (in case of respiratory distress) and fluid resuscitation (in case of tissue hypoperfusion)
Rate of evidence-based interventions initiated before hospital admission in study patients referred to from regional dispensaries | baseline
  Evidenced based interventions are defined as initiation of antimicrobials, surgical source control (if applicable), oxygen administration (in case of respiratory distress) and fluid resuscitation (in case of tissue hypoperfusion)
Rate of pre-defined adverse events | Twenty-four hours after hospital admission
Rate of evidence-based interventions performed during the first 6 hours after hospital admission before and after the implementation of a 'Sepsis First Aid' kit | Six hours after hospital admission
  Evidenced based interventions are defined as initiation of antimicrobials, surgical source control (if applicable), oxygen administration (in case of respiratory distress) and fluid resuscitation (in case of tissue hypoperfusion)
Rate of correct answers of a test on knowledge about acute infectious diseases before and after the focused educational training | 1 hour before and 1 hour after the focused educational training course

CONTACTS AND LOCATIONS:
Overall Officials: Chris Farmer, MD, Study Chair — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urayeneza O, Mujyarugamba P, Rukemba Z, Nyiringabo V, Ntihinyurwa P, Baelani JI, Kwizera A, Bagenda D, Mer M, Musa N, Hoffman JT, Mudgapalli A, Porter AM, Kissoon N, Ulmer H, Harmon LA, Farmer JC, Dunser MW, Patterson AJ; Sepsis in Resource-Limited Nations Workgroup of the Surviving Sepsis Campaign. Increasing Evidence-Based Interventions in Patients with Acute Infections in a Resource-Limited Setting: A Before-and-After Feasibility Trial in Gitwe, Rwanda. Crit Care Med. 2018 Aug;46(8):1357-1366. doi: 10.1097/CCM.0000000000003227. PMID 29957715
- [Derived] Urayeneza O, Mujyarugamba P, Rukemba Z, Nyiringabo V, Ntihinyurwa P, Baelani JI, Kwizera A, Bagenda D, Mer M, Musa N, Hoffman JT, Mudgapalli A, Porter AM, Kissoon N, Ulmer H, Harmon LA, Farmer JC, Dunser MW, Patterson AJ; Sepsis in Resource-Limited Nations Workgroup of the Surviving Sepsis Campaign. Increasing evidence-based interventions in patients with acute infections in a resource-limited setting: a before-and-after feasibility trial in Gitwe, Rwanda. Intensive Care Med. 2018 Sep;44(9):1436-1446. doi: 10.1007/s00134-018-5266-x. Epub 2018 Jun 28. PMID 29955924